CLINICAL TRIAL: NCT00500227
Title: Observational Study to Evaluate, in Acromegalic Patients With Disease Persistence After Surgery, Those Histopathologic, Clinical, Morphologic and Biochemical Factors Predictors of Hormonal Control Under Somatostatin Analogue Treatment
Brief Title: Predictive Factors of Response to Somatostatin Analogues in Acromegalic Patients With Persistent Disease Following Surgery
Acronym: ESPORA
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52030-728
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The objective of this study is to evaluate, in acromegalic patients with disease persistence after surgery who are treated with somatostatin analogues, the histopathological, clinical, morphological and biochemical factors which are predictive of hormonal control.

ELIGIBILITY:
Inclusion Criteria:

* Acromegalic patients with persistent disease (growth hormone ≥ 1ng/ml following oral glucose tolerance test and/or insulin like growth factor 1 above the normal range for sex and age) 3 to 6 months after transsphenoidal or transfrontal surgery

Exclusion Criteria:

* Patients not contributing enough material for a tumour histopathological study
* Patients who have received radiation therapy or will receive it during the observational study period
* Patients who are being treated, or in whom treatment is anticipated, with either a dopaminergic agonist or a growth hormone receptor antagonist
* Patients with a history of hypersensitivity to somatostatin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acromegalic patients with persistence of the disease who attend specialized visits (Endocrinologist) at the Spanish hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (30):
- Spain (30):
  - Hospital "Juan Canalejo", A Coruña
  - Hospital General Universitari d'Alacant, Alicante
  - Hospital de Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General de la Vall d´Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital "Mútua de Terrassa", Barcelona
  - Hospital Prínceps d'Espanya, Barcelona
  - Hospital Universitario de Getafe, Getafe
  - Complejo Hospitalario de León. Hospital Virgen Blanca., León
  - Complejo Hospitalario Xeral-Calde de Lugo, Lugo
  - Hospital de La Princesa, Madrid
  - Hospital "Ramón y Cajal", Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico de Madrid, Madrid
  - Hospital Universitario "12 de Octubre", Madrid
  - Hospital Universitario "La Paz", Madrid
  - Complexo Hospitalario de Orense, Ourense
  - Hospital "Son Dureta", Palma de Mallorca
  - Hospital de Navarra, Pamplona
  - Hospital Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital "Marqués de Valdecilla", Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital "Joan XXIII", Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Complejo Hospitalario Xeral-Cies de Vigo, Vigo
  - Hospital "Miguel Servet", Zaragoza
  - Hospital Clínico Universitario "Lozano Blesa", Zaragoza